CLINICAL TRIAL: NCT00475826
Title: Evaluation of Chylomicrons Metabolism in Sub-Clinical Atherosclerosis in Patients Whit Heterozigous Familial Hypercholesterolemia (FH) Treated With Statin Plus Ezetimibe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 1067/06
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2007-05

CONDITIONS: Heterozigous Familial Hypercholesterolemia
Keywords: Heterozigous Familial Hypercholesterolemia; Sub-clinical atherosclerosis; Chylomicrons metabolism; Statin plus ezetimibe; Coronary artery calcification
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Statins and Ezetimibe

SUMMARY:
Study Title: Evaluation of chylomicrons metabolism in sub-clinical atherosclerosis in patients whit Heterozigous Familial Hypercholesterolemia (FH) treated with statin plus ezetimibe.

Background:

Coronary artery calcification (CAC) is a marker of sub-clinical coronary atherosclerosis which correlates with higher risk of clinical events. It was already demonstrated that CAC is more prevalent in patients with FH compared with normal individuals. A number of studies demonstrated that plasmatic removal of chylomicrons is defective in patients with atherosclerosis. Despite the fact that is still controversial whether this impairment occurs in patients with HF when compared to normal controls, the kinetics of chylomicrons has not been studied in HF patients with and without atherosclerosis and more important, it is not clear if those changes may be observed in the sub-clinical disease, as reported for CAC in asymptomatic individuals.

Previous studies have demonstrated the inverse correlation among LDL-C levels and the removal of remnants chylomicrons using artificial chylomicrons technique. It is also well known that high doses of more potent statins are more effective to remove chylomicrons from the plasma due to better expression of LDL-C receptors through plasma LDL-C reduction. It was not evaluated yet if the association of ezetimibe and statin, enhancing LDL-C receptors expression in the liver would enhance the efficacy of the monotherapy with statins to remove artificial chylomicrons in patients with HF.

Study design:

Open, randomized, single-blinded study in which twenty six outpatients from the Lipids Clinical Unit at the Heart Institute (INCOR), University of São Paulo, previously diagnosed with FH according to US MED PED criteria, without history of CD and a CAC evaluation by MSCT (Multiple Sensors Computed Tomography) in the previous year will be compared to 26 control individuals matched by age and sex collected from the database of the Lipids Metabolism Laboratory.

Patients will be randomized to receive simvastatin 40 mg as monotherapy or in combination with ezetimibe 10 mg and will undergoing three kinetics studies to demonstrate the effects of simvastatin 40 mg on the kinetics of the chylomicrons along with other laboratorial dosages ( lipid fractions, hepatic enzymes and CK).

The primary endpoint of this study is to evaluate if there is any correlation among the reduction of the plasma clearance of chylomicrons by the artificial chylomicrons technique and the presence of sub-clinical atherosclerosis; the secondary endpoint is to evaluate if ezetimibe/simvastatin enhances the effects of simvastatin alone in the removal of chylomicrons in patients with HF.

ELIGIBILITY:
Inclusion Criteria:

* Heterozigous Familial Hypercholesterolemia patients
* Age 18 to 70
* Male and Female
* Coronary artery calcification

Exclusion Criteria:

* Coronary artery disease
* Cerebrovascular disease
* Diabetes Mellitus
* Heart Failure Class III-IV
* Thyroid disease
* Peripheral Artery disease
* Pregnancy, women without anticonceptive method
* Kidney disease or calcium disturbs
* Thoracic Cancer
* Use of Beta Blockers, diuretics, glucocorticoids ,hormone replacement therapy except oral anticonception
* Use of lipid lowering drugs for the last six weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-04

PRIMARY OUTCOMES:
Evaluate if there is any correlation among the reduction of the plasma clearance of chylomicrons by the artificial chylomicrons technique and the presence of sub-clinical atherosclerosis | Five months

SECONDARY OUTCOMES:
Evaluate if ezetimibe/simvastatin enhances the effects of simvastatin alone in the removal of chylomicrons in patients with HF. | Five Months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Alcova Nogueira, MD, Principal Investigator — Heart Institute-Universaty Of Sao Paulo
Locations (1):
- Heart Institute, São Paulo, São Paulo, Brazil